CLINICAL TRIAL: NCT04423549
Title: Predictive Value of a mRNA Signature and Liquid Biopsy in Diffuse Large B Cell Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Chief physician, Sun Yat-sen University
Other Study IDs: B2020-034
Record Dates: First submitted 2020-06-07; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- tested group
- controlled group

SUMMARY:
The purpose of this study is to determine the predictive value of a mRNA signature and liquid biopsy in patients with Diffuse Large B cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* biopsy proved Diffuse Large B cell Lymphoma
* newly diagnosed between 2000-01 and 2015-12

Exclusion Criteria:

* patients with biopsy samples unavailable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5-years

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Universitiy Cancer Center, Sun Yat-Sen University,, Guangzhou, China